CLINICAL TRIAL: NCT03124095
Title: Effects of Combined Training on Quality of Life, Neuromuscular and Cardiorespiratory Parameters in Patients Who Have Completed the Primary Treatment for Breast Cancer: a Randomized Clinical Trial
Brief Title: Combined Training Intervention for Women Who Underwent Primary Treatment for Breast Cancer
Acronym: +Vida
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Stephanie Santana Pinto, PhD, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: +Vida-Breast cancer
Record Dates: First submitted 2017-04-11; First posted 2017-04-21 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Breast Neoplasm
Keywords: physical exercise; combined training; physical activity; physical fitness
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combined Exercise Group (Experimental): The subjects of the combined training group will undergo the intervention three times a week for eight weeks. The combined group will carry out both resistance and aerobic exercises in the same session. The resistance training will be comprised by ten exercises which will alternate body segments with maximum repetitions in the first set and the lower limit of the repetitions interval in the next sets. Along the training, the number of series will be increased whereas the number of repetitions will be decreased. The intensity of the aerobic exercises will be based on the percentage of the heart rate of the anaerobic threshold on the first weeks and on the speed of the anaerobic and aerobic threshold on the last weeks
  Interventions: Behavioral: Combined exercise Group
- Control Group (No Intervention): The control group will be advised not to change their health habits. After the intervention they will be invited to participate in a physical exercise program.

INTERVENTIONS:
Behavioral: Combined exercise Group — The subjects of the combined training group will undergo the intervention three times a week for eight weeks. The combined group will carry out both resistance and aerobic exercises in the same session. The resistance training will be comprised by ten exercises which will alternate body segments with maximum repetitions in the first set and the lower limit of the repetitions interval in the next sets. Along the training, the number of series will be increased whereas the number of repetitions will be decreased. The intensity of the aerobic exercises will be based on the percentage of the heart rate of the anaerobic threshold on the first weeks and on the speed of the anaerobic and aerobic threshold on the last weeks
  Arms: Combined Exercise Group

SUMMARY:
The aim of the present study is analyze the effects of combined training program (resistance and aerobics) in comparison with a non-training group on quality of life, as well as on neuromuscular and cardiorespiratory parameters in breast cancer patients in stages one to three who have finished their treatment, such as surgery, chemotherapy and radiotherapy. Therefore, 42 women will be randomly divided into two groups: combined training group and control group. The subjects of the combined training group will undergo the intervention three times a week for eight weeks. The combined group will carry out both resistance and aerobic exercises in the same session. The resistance training will be comprised by ten exercises which will alternate body segments with maximum repetitions in the first set and the lower limit of the repetitions interval in the next sets. Along the training, the number of series will be increased whereas the number of repetitions will be decreased. The intensity of the aerobic exercises will be based on the percentage of the heart rate of the anaerobic threshold on the first weeks and on the speed of the anaerobic and aerobic threshold on the last weeks. Before and after the intervention, there will be evaluation of maximal dynamic strength of knee extensors and elbow flexors, maximum voluntary isometric contraction of knee extensors, maximum muscular activity of vastus lateralis and rectus femoris, muscle thickness of knee extensors, peak oxygen uptake and ventilatory threshold, quality of life and cancer-related fatigue. Data will be analyzed by Generalized Estimating Equations (GEE) and Bonferroni's post-hoc (α=0,05), including both protocol and intention to treat.

DETAILED DESCRIPTION:
According to the World Health Organization, breast cancer is the most common one among women, both in developed and developing countries. It accounts for 23% of all breast cancer cases worldwide whereas, in Brazil, it represents 25% of new cases per year. However, its mortality rate has increasingly decreased due to advances in screening protocols, diagnoses and treatment in the last decades. Even so, breast cancer and its treatment might cause psychological and physiological side effects that can affect patients' quality of life.

There is evidence that increase in physical activity generates important physical and psychological benefits to patients with cancer. Studies with breast cancer survivors have shown that the fact that the patients become physically active after the diagnosis leads to a 24-67% decrease in total death risk and 50-53% decrease in death related to breast cancer, by comparison with sedentary patients.

Reviews, systematic reviews and metaanalysis of studies that investigated the effects of interventions with physical exercise programs on health outcomes in breast cancer survivors showed the benefits brought to these patients by exercise. However, these reviews have also called the attention of the scientific community regarding the need to standardize measures of outcomes and intervention methods of evaluation since variations found in the studies make it difficult to reach definite conclusions. Furthermore, type, frequency, intensity and duration of exercise sessions to reach beneficial effects on important health parameters for breast cancer have not been well established yet. Therefore, this study aims at analyzing the effects of combined training program (resistance and aerobics), in comparison with a non-training group, on quality of life, as well as on neuromuscular and cardiorespiratory parameters in breast cancer patients in stages one to three who have finished their treatment, such as surgery, chemotherapy and radiotherapy.

Methodology: This trail will be carried out with women with histological confirmed breast cancer who have already completed the primary treatment for breast cancer (including surgery, radiation therapy and chemotherapy) from 6 months to 5 years but keep on hormone therapy. After baseline assessments, the eligible participants will be randomized to the combined exercise group or control non-exercising group. The combined exercise group will follow an eight week exercising program, which consists of three weekly exercise sessions. Each session will last around 60 minutes and will include strength training (with machines and elastic bands) and aerobic exercises on treadmills. Workouts will be guided and supervised by previously trained physical education professionals and physiotherapists. The strength training will comprise nine exercises, which will alternate body segments with maximum repetitions in the first set and the inferior limit of repetitions in the second set. Along the training, the number of series will increase whereas the number of repetitions will decrease. The intensity of the aerobic exercises will be based on the percentage of cardiac frequency of anaerobic threshold. All exercise sessions will take place at the Physical Education School at the Pelotas Federal University, located in Pelotas, Rio Grande do Sul, Brazil.

ELIGIBILITY:
Inclusion Criteria:

Volunteer women above 18 years old with histological confirmed breast cancer in stages I-IIIA who have finished their treatment, such as surgery, chemotherapy and radiotherapy.

Exclusion Criteria:

* Cardiovascular disease (except hypertension controlled by medication);
* Metastatic disease or active regional locus;
* Physical or psychiatric impairments for exercise;
* Severe nausea;
* Anorexia;
* Participation in exercise more than 75 minutes/week

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-09; Primary Completion 2017-11-26 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory Fitness evaluation change after 8 weeks | Testing of VO2peak change - Baseline and 8 week
  We created a protocol on the treadmill to determine the peak oxygen uptake change(VO2peak), the first ventilatory threshold and the second ventilatory threshold. The protocol consists in 1-minute stages. The initial speed is 1.86 miles per hour. In each stage, the speed increases 0.3 miles per hour and every 2 stages, the treadmill inclination increases 1%. The test is interrupted when the subject indicates exhaustion. The respiratory gases will be collected through a portable gas analyzer (VO2000, MedGraphics, Ann Arbor, USA).
  The maximum value of VO2 , closed to exhaustion will be considered the VO2peak. The fist and the second ventilatory threshold will be determined by the ventilation versus intensity curve and confirmed by the O2 and Carbon dioxide ventilatory equivalents by two independent physiologists in a visual inspection.

SECONDARY OUTCOMES:
Quality of Life change after 8 weeks (Score) | Baseline and 8 week
  Functional Assessment of Cancer Therapy- Breast.
Maximal dynamic strength change after 8 weeks (kg) | Baseline and 8 week
  1- maximum repetition of knee extensors
maximum voluntary isometric contraction of knee extensors change after 8 weeks | Baseline and 8 week
  load cell
Cancer related fatigue change after 8 weeks | Baseline and 8 week
  Piper Fatigue Scale
muscle thickness of knee extensors change after 8 weeks | Baseline and 8 week
  ultrasound image
maximum muscular activity of vastus lateralis and rectus femoris change after 8 weeks | baseline and 8 weeks
  electromyography

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Education School, Pelotas, Rio Grande do Sul, Brazil